CLINICAL TRIAL: NCT00727454
Title: Effects of Continuous Positive Airway Pressure on Heart Remodeling in Patients With Obstructive Sleep Apnea: A Randomized Study With Cardiovascular Magnetic Resonance Imaging
Brief Title: Effects of Continuous Positive Airway Pressure (CPAP) in Heart Remodeling by Magnetic Resonance Imaging (MRI)
Acronym: OSA-MRI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty of recruiting patients and cost limitations.
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Luciano F Drager, Luciano F. Drager, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3163/08/79
Record Dates: First submitted 2008-07-28; First posted 2008-08-04 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; CPAP; Heart remodeling; Cardiovascular disease; MRI
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Control (Placebo Comparator): No treatment
  Interventions: Device: No treatment
- 2 CPAP (Experimental): Continuous Positive Airway Pressure (CPAP) - REMStar Pro with C-Flex; Respironics, Inc., Murrysville, PA
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — Continuous Positive Airway Pressure (CPAP) during sleep for 3 months.
  Other Names: CPAP REMStar Pro with C-Flex; Respironics, Inc.
  Arms: 2 CPAP
Device: No treatment — No treatment
  Arms: 1 Control

SUMMARY:
Obstructive sleep apnea (OSA) is independently associated with important heart remodeling that further contributes to overt heart failure. Recent evidences using echocardiogram suggested that continuous positive airway pressure (CPAP) has beneficial effects mainly on left ventricle parameters. However, the evidences regarding the right ventricle are scanty. In addition, no previous studies evaluated morphological and functional characteristics in OSA by magnetic resonance imaging (MRI) as well as the impact of CPAP.

DETAILED DESCRIPTION:
The patients will be recruited from the Sleep Laboratory, Heart Institute (InCor), University of São Paulo Medical School. Male adults with a sleep study within 1 month showing severe OSA (>30 events of apnea and hypopnea per hour of sleep) and naive to treatment will be considered for the study. Age and body mass index matched controls will be recruited from the hospital staff and their relatives. All volunteers will be previously screening for the risk of OSA with Berlin Questionnaire. To minimize confounding risk factors, we will exclude subjects older than 60 years and those with a body mass index (BMI) >40 kg/m2, diabetes mellitus, hypertension, cerebrovascular disease, valvular heart disease, renal failure, current or past smoking history, and chronic use of any medication. Hypertension will be excluded after 3 or more normal blood pressure values (<140/90mm Hg) obtained on separate occasions with a conventional mercury sphygmomanometer.

Sleep Study. All participants will perform a standard overnight polysomnography. Apnea will be defined as complete cessation of airflow for at least 10 seconds, associated with oxygen desaturation of 3%. Hypopnea will be defined as a significant reduction (>50%) in respiratory signals for at least 10 seconds associated with oxygen desaturation of 3%. The apnea-hypopnea index will be calculated as the total number of respiratory events (apneas plus hypopneas) per hour of sleep. Normal values will be considered when the apnea-hypopnea index will be <5events/hour.

The participants will be randomly assigned to no treatment (control) or treatment with CPAP for 3 months, according to a computer-generated list of random numbers. At baseline and after 3 months, the participants will be submitted to cardiac MRI.

Magnetic resonance imaging methods. Participants will perform MRI examination on 1.5 - T GE CV/i system. Short and long-axis of the heart will be obtained during breath-hold and triggered on electrocardiogram pulse sequences. The first sequence will be a gradient-echo (steady-sate free procession) to assess left ventricular (LV) and right ventricular (RV) morphology and function. The second sequence will be an inversion-recovery prepared gradient-echo to obtain MDE (10 to 20 minutes after intravenous bolus of 0.2 mmol/Kg of gadolinium-based contrast). We will use the following parameters: repetition time 3.9/7.1ms, echo time 1.7/3.1 ms, flip angle 45º/20º, cardiac phases 20/1, views per segment 8/16 to 32, matrix 256 x 128/256 x 192, slice thickness 8/8mm, gap between slices 2/2mm and field of view 32 to 38/32 to 38 cm, inversion time none/150 to 250 ms, receiver bandwidth 125/31,25 kHz, number of excitations 1/2.

Blood Samples. Venous blood will be collected from all participants between 8 and 10 AM for the measurement of glucose, total cholesterol, low-density lipoprotein, high-density lipoprotein, and red blood cell count.

24-hour blood pressure monitoring. All participants will be submitted to a 24-hour blood pressure monitoring with a SpaceLabs device (model 90207).

ELIGIBILITY:
Inclusion Criteria:

* Patients free of comorbidities with severe Obstructive Sleep Apnea by polysomnography.
* Healthy volunteers (no obstructive sleep apnea and no comorbidities) matched for age, sex and body mass index.

Exclusion Criteria:

* Subjects older than 60 years
* Body mass index (BMI) >40 kg/m2
* Diabetes mellitus
* Hypertension
* Cerebrovascular disease
* Valvular heart disease
* Renal failure
* Current or past smoking history
* Chronic use of any medication

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-07; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Right ventricle parameters: size and function. | Baseline and after 3 months.

SECONDARY OUTCOMES:
Left Ventricle parameters: size and function | Baseline and after 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano F Drager, MD, PhD, Principal Investigator — Hypertension Unit, Heart Institute (InCor)
Locations (2):
- Brazil (2):
  - Heart Institute (InCor) - University of São Paulo Medical School, São Paulo, São Paulo
  - Heart Institute (InCor), São Paulo, São Paulo